CLINICAL TRIAL: NCT01916772
Title: Natural Hisotry of Cherubism Observational Study
Brief Title: Natural History of Cherubism Observational Study
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: CCFO7256
Record Dates: First submitted 2013-07-25; First posted 2013-08-06 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Cherubism
Keywords: cherubism; bone tumors
MeSH Terms: conditions — Cherubism; Bone Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We may take blood or skin samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cherubism patients: no interventions
  Interventions: Other: no interventions

INTERVENTIONS:
Other: no interventions — no interventions

SUMMARY:
To observe the natural history of cherubism.

DETAILED DESCRIPTION:
The investigators will take a history and examine patients with cherubism to determine the natural history of the disease. The investigators also may take skin or blood samples (IRB approved 7256) from patients to learn more about this disorder.

ELIGIBILITY:
Inclusion Criteria:

patients with cherubism

Exclusion Criteria:

patients without cherubism

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We will see patients with cherubism
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2013-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Disease progression | 10 years
  We will take a history and examine patients with cherubism and look for disease progression.

SECONDARY OUTCOMES:
patient growth | 10 years
  We will measure height and weight
bone abnormalities | 10 years
  We will take panorex radiographs.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lietman, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Background] Lietman SA, Kalinchinko N, Deng X, Kohanski R, Levine MA. Identification of a novel mutation of SH3BP2 in cherubism and demonstration that SH3BP2 mutations lead to increased NFAT activation. Hum Mutat. 2006 Jul;27(7):717-8. doi: 10.1002/humu.9433. PMID 16786512
- [Background] Fan C, Gaivin RJ, Marth TA, Willard B, Levine MA, Lietman SA. Cloning and characterization of the human SH3BP2 promoter. Biochem Biophys Res Commun. 2012 Aug 17;425(1):25-32. doi: 10.1016/j.bbrc.2012.07.043. Epub 2012 Jul 17. PMID 22820184
- [Background] Reichenberger EJ, Levine MA, Olsen BR, Papadaki ME, Lietman SA. The role of SH3BP2 in the pathophysiology of cherubism. Orphanet J Rare Dis. 2012 May 24;7 Suppl 1(Suppl 1):S5. doi: 10.1186/1750-1172-7-S1-S5. Epub 2012 May 24. PMID 22640988